CLINICAL TRIAL: NCT05590273
Title: Forgotten Voices: Addressing Unmet Needs in Brain Tumor Caregivers (AIM 2)
Brief Title: Forgotten Voices: Addressing Unmet Needs in Brain Tumor Caregivers
Acronym: AIM 2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient caregiver participation
Sponsor: Virginia Commonwealth University (Other)
Collaborators: American Psychological Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-22-19366; HM20024428 (Other: Virginia Commonwealth University)
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Caregivers; Neuro-Oncology; Brain Cancer
Keywords: CALM
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: This study has been designed in accordance with the NIH Science of Behavior Change ORBIT model for developing behavioral interventions and represents a Phase Ia Define Trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Proof-of-concept trial (Experimental): Inform CALM adaptations for caregivers of patients with brain cancer.
  Interventions: Behavioral: CALM Therapy

INTERVENTIONS:
Behavioral: CALM Therapy — The CALM intervention includes 3 to 6 individual therapy Zoom teletherapy sessions, each approximately 50-60 minutes in length biweekly, delivered over 3 months. Participants (caregivers) will be asked to complete self-report surveys of behavioral and psychological variables surveys at the following timepoints:
  Within one week before initiating the CALM intervention therapy (baseline) and immediately after the program (post-intervention)
  In addition, after each intervention session, participants will complete a brief post-session survey to assess acceptability of CALM session components.
  Lastly, participants will complete an exit interview immediately following the end of the intervention.

SUMMARY:
To conduct a mixed-method Phase Ia Define Trial of caregivers' participation in CALM therapy with post-session surveys and individual exit interviews in order to evaluate suitability and adapt the CALM intervention to the needs of caregivers in neuro-oncology.

DETAILED DESCRIPTION:
Exploring caregivers' experiences of CALM intervention will inform more effective, targeted, supportive care for this traditionally underserved group in need of emotional support. We will use the data from this study to adapt the CALM intervention to the specific needs of caregivers in neuro-oncology

ELIGIBILITY:
Inclusion Criteria:

* Caregiver participants must be the caregiver of a brain cancer patient who is currently enrolled in DoD CA200896 (IRBHM20022755)
* Fluent in English
* Willing and able to attend a minimum of 3 CALM sessions via telehealth
* A caregiver is defined as the primary person who provides ongoing support to the brain cancer patient; it is not necessary that the caregiver lives with the patient or is related
* Patient participants must have enrolled in the linked HM20022755 study

Exclusion Criteria:

* Person does not consider themselves to be a caregiver of the patient
* Caregiver does not have a loved one (patient diagnosed with brain cancer) enrolled in DoDCA200896 (IRB HM20022755)
* Caregiver does not speak English
* Caregiver is unable to provide consent
* Caregiver does not have access to telehealth
* Caregiver is under the age of 18
* Professional caregivers who received financial compensation for their services are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Evaluate suitability of the CALM intervention to the needs of caregivers in neuro-oncology by measuring caregiver satisfaction. | 3 months
  Utilizing post-session surveys, determine caregiver satisfaction (5-point Likert Scale) with 1) topic applicability; 2) perceived benefit of session; 3) comfort with interventionist(s); 4) overall satisfaction and 5) likelihood of recommending the program to others. Higher scores represent greater caregiver satisfaction with the CALM intervention.
Evaluate suitability of the CALM intervention to the needs of caregivers in neuro-oncology by measuring caregivers' recommendations to the content and format of the intervention during an exit-interview. | 3 months
  Caregivers will be asked a number of open-ended questions about their recommendations to CALM during a semi-structured exit interview. Exit interviews will be audio recorded and transcribed verbatim. A co- investigator and a second independent coder will separately review each transcript to identify common themes and develop a coding framework of free responses. All results will be reviewed for agreement and comparison to the raw data, and discrepancies will be resolved through discussion with the PI until reliability is reached (Kappa>.80).

CONTACTS AND LOCATIONS:
Overall Officials: Ashlee R Loughan, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-09-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT05590273/ICF_000.pdf